CLINICAL TRIAL: NCT04667377
Title: A Phase II, Randomized, Double Blind, Parallel Group,46 Weeks Dose-finding Study of BI 456906 Administered Once Weekly Subcutaneously Compared With Placebo in Patients With Obesity or Overweight
Brief Title: A Study to Test Whether Different Doses of BI 456906 Help People With Overweight or Obesity to Lose Weight
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1404-0036; 2020-002479-37 (EudraCT Number)
Record Dates: First submitted 2020-12-08; First posted 2020-12-14 (Actual); Results first posted 2023-11-02 (Actual); Last update posted 2023-11-02 (Actual); Status verified 2023-10

CONDITIONS: Obesity
MeSH Terms: conditions — Obesity | interventions — BI 456906

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- 0.6 mg BI 456906 (Experimental)
  Interventions: Drug: BI 456906
- Placebo group (Placebo Comparator)
  Interventions: Drug: Placebo
- 2.4 mg BI456906 (Experimental)
  Interventions: Drug: BI 456906
- 3.6 mg BI 456906 (Experimental)
  Interventions: Drug: BI 456906
- 4.8 mg BI 456906 (Experimental)
  Interventions: Drug: BI 456906

INTERVENTIONS:
Drug: BI 456906 — BI 456906
  Other Names: Survodutide
  Arms: 0.6 mg BI 456906; 2.4 mg BI456906; 3.6 mg BI 456906; 4.8 mg BI 456906
Drug: Placebo — Placebo
  Arms: Placebo group

SUMMARY:
This study is open to adults, aged 18 to 75 years, with overweight or obesity. People with body mass index (BMI) of 27 or higher to join the study. People who have diabetes cannot participate. The purpose of this study is to find out whether a medicine called BI 456906 helps people lose weight.

Participants are put into 5 groups by chance. 4 groups get different doses of BI 456906. The fifth group gets placebo. Participants get BI 456906 or placebo as injections under the skin once a week. Placebo injections look like BI 456906 injections but do not contain any medicine.

Participants are in the study for about a year. During this time, there are about 20 in-person visits to the study site. At the study site visits, doctors measure participants' body weight. Results are compared between the BI 456906 groups and the placebo group. The doctors also regularly check the general health of the participants.

ELIGIBILITY:
Inclusion Criteria:

* Adult ≥ 18 years and < 75 years of age at screening
* Signed and dated written informed consent in accordance with ICH-GCP and local legislation prior to admission to the trial.
* Obesity or Overweight defined as BMI ≥27 kg/m2 at screening
* A minimum absolute body weight of 70 kg for females and 80 kg for males at screening
* Male or female participants. Women of childbearing potential (WOCBP)1 must be willing and able to use two forms of effective contraception where at least one form is highly effective methods of birth control per ICH M3 (R2) that result in a low failure rate of less than 1% per year when used consistently and correctly. A list of contraception methods meeting these criteria is provided in the patient information.
* Patients must have undergone at least one previous unsuccessful nonsurgical weight-loss attempt per investigator's judgement

Exclusion criteria:

* Body weight change of over +/- 5% or more in the past 12 weeks prior to randomization. There must be documentation of weight in the past 12 weeks before randomization.
* Obesity induced by an endocrinologic disorder (i.e. Cushing Syndrome, hypogonadism, growh hormone deficiency. However, well controlled hypothyroidism, polycystic ovarian disease are still allowed)
* A HbA1c ≥ 6.5% at screening or diagnosed with type 1 or type 2 diabetes mellitus
* Exposure to Glucagon like peptide-1 receptor agonist (GLP-1Ra) based therapies within three months prior to screening
* Any suicidal behaviour in the past 2 years, any suicidal ideation of type 4 or 5 in the Columbia-Suicide Severity Rating Scale (CSSRS) within 3 months before screening, or during screening period
* History of major depressive disorder within 2 years before randomization
* Major depressive symptoms (defined as a screening Patient Health Questionnaire-9 [PHQ-9] score ≥15) at screening and/or during screening period
* Diseases of the central nervous system (including but not limited to any kind of seizures or stroke), and other relevant neurological or psychiatric disorders at screening
* Chronic or relevant acute infections (including but not limited to respiratory tract infections, urinary tract infection, bladder infection, enterocolitis, abscess, tuberculosis, meningitis, influenza, Epstein-Barr virus, HIV/AIDS, and hepatitis B or C, and severe acute respiratory syndrome coronavirus type 19 (SARS CoV-2) (as confirmed by Polychain reaction (PCR) test)), within 2 weeks from screening or during screening.
* Further exclusion criteria apply

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 387 (Actual)
Dates: Start 2021-03-08 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-10-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (43):
- United States (10):
  - Diablo Clinical Research, Walnut Creek, California
  - L-MARC Research Center, Louisville, Kentucky
  - Lucas Research, Inc., Morehead City, North Carolina
  - PMG Research of Wilmington, LLC, Wilmington, North Carolina
  - Valley Weight Loss Clinic, Fargo, North Dakota
  - Velocity Clinical Research, Inc., Cleveland, Ohio
  - TLM Medical Services, LLC, Columbia, South Carolina
  - Coastal Carolina Research Center, North Charleston, South Carolina
  - Washington Center for Weight Management and Research, Inc., Arlington, Virginia
  - Allegiance Research Specialists, Wauwatosa, Wisconsin
- Australia (5):
  - The Boden Initiative, Camperdown, New South Wales
  - Nepean Hospital, Kingswood, New South Wales
  - Royal Adelaide Hospital, Adelaide, South Australia
  - Eastern Clinical Research Unit, East Ringwood, Victoria
  - Austin Health, Heidelberg, Victoria
- UZ Leuven, Leuven, Belgium
- Canada (5):
  - Joanne F Liutkus Medicine Professional Corporation, Cambridge, Ontario
  - Bluewater Clinical Research, Sarnia, Ontario
  - Canadian Phase Onward Inc., Toronto, Ontario
  - LMC Clinical Research Inc. (Bayview), Toronto, Ontario
  - Recherche GCP Research, Montreal, Quebec
- China (4):
  - Beijing Chao-Yang Hospital, Beijing
  - Beijing Luhe Hospital Capital Medical University, Beijing
  - The First Hospital of Jilin University, Changchun
  - Wuhan Union Hospital, Wuhan
- Germany (2):
  - Klinische Forschung Berlin GbR, Berlin
  - Universitätsklinikum Carl Gustav Carus Dresden, Dresden
- Netherlands (4):
  - EB Flevoresearch, Almere Stad
  - PT & R, Beek
  - Franciscus Gasthuis, Rotterdam
  - Albert SchweitzerZiekenhuis, Zwijndrecht
- New Zealand (2):
  - Optimal Clinical Trials, Auckland
  - P3 Research, Newtown Wellington NZ
- Poland (2):
  - Salvia Lekston I Madej Sp. J., Katowice
  - Metabolic Health Center Pawel Bogdanski, Poznan
- South Korea (3):
  - Seoul National University Bundang Hospital, Seongnam
  - Kyung Hee University Hospital at Gangdong, Seoul
  - The Catholic University of Korea, Yeouido St.Mary's Hospital, Seoul
- Sweden (3):
  - Ladulaas Kliniska Studier, Borås
  - Forskningsenheten Carlanderska, Gothenburg
  - Akademiska sjukhuset, Uppsala
- United Kingdom (2):
  - Waterloo Medical Centre, Blackpool
  - Clifton Medical Centre, Rotherham, Rotherham

IPD SHARING:
Plan to Share IPD: Yes
After the study is completed and the primary manuscript is accepted for publishing, researchers can use this following link https://www.mystudywindow.com/msw/datasharing to request access to the clinical study documents regarding this study, and upon a signed "Document Sharing Agreement".
  Also, Researchers can use the following link https://www.mystudywindow.com/msw/datasharing to find information in order to request access to the clinical study data, for this and other listed studies, after the submission of a research proposal and according to the terms outlined in the website.
  The data shared are the raw clinical study data sets.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After all regulatory activities are completed in the US and EU for the product and indication, and after the primary manuscript has been accepted for publication.
Access Criteria: For study documents - upon signing of a 'Document Sharing Agreement'. For study data - 1. after the submission and approval of the research proposal (checks will be performed by both the independent review panel and the sponsor, including checking that the planned analysis does not compete with sponsor's publication plan); 2. and upon signing of a 'Data Sharing Agreement'.
URL: https://www.mystudywindow.com/msw/datasharing

REFERENCES:
- [Derived] le Roux CW, Steen O, Lucas KJ, Startseva E, Unseld A, Hussain SA, Hennige AM. Subgroup analysis by sex and baseline BMI in people with a BMI >/=27 kg/m2 in the phase 2 trial of survodutide, a glucagon/GLP-1 receptor dual agonist. Diabetes Obes Metab. 2025 Apr;27(4):1773-1782. doi: 10.1111/dom.16167. Epub 2025 Jan 16. PMID 39821928
- [Derived] le Roux CW, Steen O, Lucas KJ, Startseva E, Unseld A, Hennige AM. Glucagon and GLP-1 receptor dual agonist survodutide for obesity: a randomised, double-blind, placebo-controlled, dose-finding phase 2 trial. Lancet Diabetes Endocrinol. 2024 Mar;12(3):162-173. doi: 10.1016/S2213-8587(23)00356-X. Epub 2024 Feb 5. PMID 38330987
- See also: Related Info — https://www.mystudywindow.com/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a randomised, double-blinded, parallel-design, placebo-controlled, multi-national, and multi-centre study with four different BI 456906 maintenance doses (ranging from 0.6 mg/week to 4.8 mg/week) in patients with obesity or overweight (body mass index (BMI) >=27 kg/m^2), and without diabetes mellitus.
Pre-assignment Details: All subjects were screened for eligibility prior to participation in the trial. Subjects attended a specialist site which ensured that they (the subjects) strictly met all inclusion and none of the exclusion criteria. Subjects were not to be allocated to a treatment group if any of the entry criteria were violated.
Groups:
- 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation): Participants with obesity or overweight were administered a solution for injection of BI 456906, by a weekly subcutaneous injection of two syringes (0.5 mL filling volume per syringe) on the same injection day, of 0.3 mg on Week 1 and 2, and 0.6 mg on Week 3 to Week 20 (dose escalation phase, with fixed dose escalation from Week 1 to Week 10 and flexible dose escalation from Week 11 to Week 20).
  From Week 21 to Week 46 (maintenance dosing phase) participants stayed on the dose of 0.6 mg BI 456906.
  Participant not tolerating the assigned dose escalation schedule due to gastrointestinal adverse events had the option of dose adjustment during the flexible part of the dose escalation phase (Week 11 - 20) which could lead to a maintenance dose lower than the dose the participant was randomised to.
- 2.4 mg BI 456906 - Planned Maintenance Treatment: Participants with obesity or overweight were administered a solution for injection of BI 456906, by a weekly subcutaneous injection of two syringes (0.5 mL filling volume per syringe) on the same injection day, of 0.3 mg on Week 1 and Week 2, 0.6 mg on Week 3 and Week 4, 0.9 mg on Week 5 and Week 6, 1.2 mg on Week 7 to Week 10, 1.8 mg on Week 11 to Week 14 and 2.4 mg on Week 15 to Week 20 (dose escalation phase, with fixed dose escalation from Week 1 to Week 10 and flexible dose escalation from Week 11 to Week 20). From Week 21 to Week 46 (maintenance dosing phase) participants stayed on the dose of 2.4 mg BI 456906.
  Participant not tolerating the assigned dose escalation schedule due to gastrointestinal adverse events had the option of dose adjustment during the flexible part of the dose escalation phase (Week 11 - 20) which could lead to a maintenance dose lower than the dose the participant was randomised to.
- 3.6 mg BI 456906 - Planned Maintenance Treatment: Participants with obesity or overweight were administered a solution for injection of BI 456906, by a weekly subcutaneous injection of two syringes (0.5 mL filling volume per syringe) on the same injection day, of 0.3 mg on Week 1 and Week 2, 0.6 mg on Week 3 and Week 4, 0.9 mg on Week 5 and Week 6, 1.2 mg on Week 7 to Week 10, 1.8 mg on Week 11 and Week 12, 2.4 mg on Week 13 and Week 14, 3.0 mg on Week 15 and Week 16, and 3.6 mg on Week 17 to Week 20 (dose escalation phase, with fixed dose escalation from Week 1 to Week 10 and flexible dose escalation from Week 11 to Week 20). From Week 21 to Week 46 (maintenance dosing phase) participants stayed on the dose of 3.6 mg BI 456906.
  Participant not tolerating the assigned dose escalation schedule due to gastrointestinal adverse events had the option of dose adjustment during the flexible part of the dose escalation phase (Week 11 - 20) which could lead to a maintenance dose lower than the dose the participant was randomised to.
- 4.8 mg BI 456906 - Planned Maintenance Treatment: Participants with obesity or overweight were administered a solution for injection of BI 456906, by a weekly subcutaneous injection of two syringes (0.5 mL filling volume per syringe) on the same injection day, of 0.3 mg on Week 1 and Week 2, 0.6 mg on Week 3 and Week 4, 0.9 mg on Week 5 and Week 6, 1.2 mg on Week 7 and Week 8, 1.8 mg on Week 9 and Week 10, 2.4 mg on Week 11 and Week 12, 3.3 mg on Week 13 and Week 14, 4.2 mg on Week 15 and Week 16, and 4.8 mg on Week 17 to Week 20 (dose escalation phase, with fixed dose escalation from Week 1 to Week 10 and flexible dose escalation from Week 11 to Week 20). From Week 21 to Week 46 (maintenance dosing phase) participants stayed on the dose of 4.8 mg BI 456906.
  Participant not tolerating the assigned dose escalation schedule due to gastrointestinal adverse events had the option of dose adjustment during the flexible part of the dose escalation phase (Week 11 - 20) which could lead to a maintenance dose lower than the dose the participant was randomised to.
- Placebo: Participants with obesity or overweight were administered a solution for injection of Placebo, by a weekly subcutaneous injection of two syringes on the same injection day, for 46 weeks.
Period: Dose Escalation Period
Arm/Group | 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) | 2.4 mg BI 456906 - Planned Maintenance Treatment | 3.6 mg BI 456906 - Planned Maintenance Treatment | 4.8 mg BI 456906 - Planned Maintenance Treatment | Placebo
Started (Randomised) | 78 | 78 | 77 | 77 | 77
Treated During Dose Escalation Period | 77 | 78 | 77 | 77 | 77
Completed (Completed = Completed trial medication) | 55 | 60 | 59 | 55 | 57
Not Completed | 23 | 18 | 18 | 22 | 20
Not completed — Other not specified below | 3 | 3 | 2 | 1 | 3
Not completed — Protocol Violation | 2 | 2 | 0 | 2 | 1
Not completed — Burden of study procedures | 2 | 1 | 1 | 1 | 5
Not completed — Change of residence | 0 | 0 | 1 | 0 | 0
Not completed — Perceived lack of efficacy | 0 | 0 | 0 | 0 | 6
Not completed — Adverse Event | 9 | 10 | 12 | 17 | 3
Not completed — Adverse event: COVID-infection | 4 | 1 | 2 | 1 | 0
Not completed — Not treated | 1 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 0 | 0 | 0 | 2
Not completed — Lost to Follow-up | 0 | 1 | 0 | 0 | 0
Period: Maintenance Period
Arm/Group | 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) | 2.4 mg BI 456906 - Planned Maintenance Treatment | 3.6 mg BI 456906 - Planned Maintenance Treatment | 4.8 mg BI 456906 - Planned Maintenance Treatment | Placebo
Started | 55 | 60 | 59 | 55 | 57
Completed (Completed = Completed trial medication) | 47 | 45 | 48 | 47 | 46
Not Completed | 8 | 15 | 11 | 8 | 11
Not completed — Perceived lack of efficacy | 0 | 2 | 1 | 0 | 1
Not completed — Adverse Event | 2 | 8 | 5 | 4 | 1
Not completed — Adverse event: COVID infection | 0 | 1 | 0 | 0 | 0
Not completed — COVID-related | 0 | 0 | 1 | 1 | 0
Not completed — Protocol Violation | 1 | 0 | 0 | 0 | 1
Not completed — Burden of study procedures | 1 | 2 | 0 | 1 | 0
Not completed — Change of residence | 0 | 1 | 0 | 0 | 1
Not completed — Missing | 1 | 0 | 0 | 0 | 0
Not completed — Other than listed above | 2 | 0 | 3 | 2 | 6
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis set (FAS): All randomised participants who received at least one dose of trial medication and who had analysable data for at least one efficacy endpoint, using planned maintenance treatment.
Groups:
- Total: Total of all reporting groups
Arm/Group | 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) | 2.4 mg BI 456906 - Planned Maintenance Treatment | 3.6 mg BI 456906 - Planned Maintenance Treatment | 4.8 mg BI 456906 - Planned Maintenance Treatment | Placebo | Total
Number analyzed (Participants) | 77 | 78 | 76 | 76 | 77 | 384
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.6 (12.6) | 49.0 (13.1) | 50.3 (11.8) | 47.6 (13.5) | 50.0 (13.5) | 48.9 (12.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 51 | 54 | 51 | 53 | 53 | 262
  Male | 26 | 24 | 25 | 23 | 24 | 122
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 2 | 6 | 5 | 17
  Not Hispanic or Latino | 74 | 77 | 74 | 70 | 72 | 367
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 0 | 1
  Asian | 8 | 9 | 9 | 7 | 7 | 40
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 1 | 1 | 2
  Black or African American | 10 | 8 | 3 | 8 | 8 | 37
  White | 59 | 60 | 63 | 59 | 60 | 301
  More than one race | 0 | 1 | 1 | 0 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Body weight at baseline [Mean (Standard Deviation); unit: Kilogram (kg)] | 106.98 (18.71) | 106.57 (22.97) | 104.68 (19.63) | 105.86 (17.39) | 104.32 (22.95) | 105.68 (20.39)

OUTCOME MEASURES:

1. Primary Outcome: Percentage Change in Body Weight From Baseline to Week 46
Description: Percentage change in body weight from baseline to Week 46 was modeled using a mixed model for repeated measures (MMRM) with fixed effects for baseline body weight as a continuous linear covariate, and treatment, gender, visit, treatment by visit interaction and baseline by visit interaction as factors, using visit (Week 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 28, 32, 36, 40, and 46) as repeated measures, an unstructured covariance matrix to model within subject measurements, adjusted mean (standard error) at Week 46 is reported. For analysis, all available post-baseline body weight measurements (on- and off-treatment) were used, except those for participants who discontinued treatment early due to COVID-19. For these participants only on-treatment values were used. That is, a hypothetical strategy was used for intercurrent event (ICE) "COVID-19 pandemic-related early treatment discontinuation", a treatment policy strategy for ICE "non-pandemic-related early treatment discontinuation".
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 28, 32, 36, 40, and 46.
Population: Full analysis set (all randomised participants who received at least one dose of study treatment and who have analysable data for at least one efficacy endpoint) using planned maintenance treatment. Number of participants analysed = Participants with available data for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Percentage change
Arm/Group | 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) | 2.4 mg BI 456906 - Planned Maintenance Treatment | 3.6 mg BI 456906 - Planned Maintenance Treatment | 4.8 mg BI 456906 - Planned Maintenance Treatment | Placebo
Number analyzed (Participants) | 76 | 78 | 76 | 76 | 77
Percentage change | -6.19 (1.07) | -12.51 (1.01) | -13.22 (1.04) | -14.94 (1.01) | -2.82 (1.06)
Statistical Analysis 1: Comparison: 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) vs 2.4 mg BI 456906 - Planned Maintenance Treatment vs 3.6 mg BI 456906 - Planned Maintenance Treatment vs 4.8 mg BI 456906 - Planned Maintenance Treatment vs Placebo; A flat vs. non-flat dose-response relationship across the 4 doses of BI 456906 and placebo was tested using the Multiple Comparison Procedure - Modelling (MCP-Mod) approach which evaluated simultaneously 5 different potential dose-response patterns (Linear, Exponential, Emax1, Emax2, Sigmoid Emax) while protecting the overall probability of type I error (one-sided alpha of 2.5%); Test type: Other — Covariate adjusted fixed effect estimates of mean percentage change in body weight at Week 46 for each treatment group with associated covariance matrix were extracted from the MMRM (including fixed effects for baseline body weight as a continuous linear covariate, and treatment, gender, visit, treatment by visit interaction and baseline by visit interaction as factors) and used as input for the MCP-Mod; p < 0.0001, MCP-Mod - Linear model fit — P-value is adjusted for multiplicity
Statistical Analysis 2: Comparison: 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) vs 2.4 mg BI 456906 - Planned Maintenance Treatment vs 3.6 mg BI 456906 - Planned Maintenance Treatment vs 4.8 mg BI 456906 - Planned Maintenance Treatment vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, MCP-Mod - Exponential model fit — P-value is adjusted for multiplicity; Model Assumption: 50% of maximum effect achieved at dose 3.6 mg
Statistical Analysis 3: Comparison: 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) vs 2.4 mg BI 456906 - Planned Maintenance Treatment vs 3.6 mg BI 456906 - Planned Maintenance Treatment vs 4.8 mg BI 456906 - Planned Maintenance Treatment vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, MCP-Mod - Emax1 model fit — P-value is adjusted for multiplicity; Model Assumption: 90% of maximum effect achieved at dose 4.8 mg
Statistical Analysis 4: Comparison: 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) vs 2.4 mg BI 456906 - Planned Maintenance Treatment vs 3.6 mg BI 456906 - Planned Maintenance Treatment vs 4.8 mg BI 456906 - Planned Maintenance Treatment vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, MCP-Mod - Emax2 model fit — P-value is adjusted for multiplicity; Model Assumption: 70% of maximum effect achieved at dose 4.8 mg
Statistical Analysis 5: Comparison: 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) vs 2.4 mg BI 456906 - Planned Maintenance Treatment vs 3.6 mg BI 456906 - Planned Maintenance Treatment vs 4.8 mg BI 456906 - Planned Maintenance Treatment vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Other — [test comment as in outcome 1, analysis 1]; p < 0.0001, MCP-Mod - Sigmoid Emax model fit — P-value is adjusted for multiplicity; Model Assumption: 50% of maximum effect achieved at dose 2.4 mg, 90% of maximum effect achieved at dose 4.8 mg
Statistical Analysis 6: Comparison: 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) vs Placebo; No formal hypotheses were tested; Test type: Other — MMRM with fixed effects for baseline body weight as a continuous linear covariate, and treatment, gender, visit, treatment by visit interaction and baseline by visit interaction as factors, using visit as repeated measures and an unstructured covariance matrix to model within subject measurements; p = 0.0257, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger approximation was used to estimate the denominator degrees of freedom; Difference of adjusted means = -3.37, 95% CI 2-sided [-6.33 to -0.41], Standard Error of Mean 1.50 — Difference was calculated as BI 456906 - placebo
Statistical Analysis 7: Comparison: 2.4 mg BI 456906 - Planned Maintenance Treatment vs Placebo; No formal hypotheses were tested; Test type: Other — [test comment as in outcome 1, analysis 6]; p < .0001, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger approximation as used to estimate the denominator degrees of freedom; Difference of adjusted means = -9.69, 95% CI 2-sided [-12.57 to -6.81], Standard Error of Mean 1.46 — Difference was calculated as BI 456906 - placebo
Statistical Analysis 8: Comparison: 3.6 mg BI 456906 - Planned Maintenance Treatment vs Placebo; No formal hypotheses were tested; Test type: Other — [test comment as in outcome 1, analysis 6]; p < .0001, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger approximation was used to estimate the denominator degrees of freedom; Difference of adjusted means = -10.40, 95% CI 2-sided [-13.32 to -7.49], Standard Error of Mean 1.48 — Difference was calculated as BI 456906 - placebo
Statistical Analysis 9: Comparison: 4.8 mg BI 456906 - Planned Maintenance Treatment vs Placebo; No formal hypotheses were tested; Test type: Other — [test comment as in outcome 1, analysis 6]; p < .0001, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger approximation will be used to estimate the denominator degrees of freedom; Difference of adjusted means = -12.12, 95% CI 2-sided [-15.00 to -9.24], Standard Error of Mean 1.46 — Difference was calculated as BI 456906 - placebo

2. Secondary Outcome: Weight Loss of ≥ 5% of Baseline Weight at Week 46
Description: Weight loss of greater than or equal to 5 percent (≥5%) of baseline weight at Week 46 (yes/no), reported as percentage of participants who achieved a weight loss of ≥5% of baseline weight at Week 46. For analysis, all available post-baseline body weight measurements (on- and off-treatment) were used, except those for participants who discontinued treatment early due to COVID-19. For these participants only on-treatment values were used. Percentages were rounded to one decimal place.
Time Frame: At baseline and at Week 46.
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) | 2.4 mg BI 456906 - Planned Maintenance Treatment | 3.6 mg BI 456906 - Planned Maintenance Treatment | 4.8 mg BI 456906 - Planned Maintenance Treatment | Placebo
Number analyzed (Participants) | 56 | 58 | 61 | 64 | 54
Percentage of participants | 60.7 | 81.0 | 82.0 | 82.8 | 25.9
Statistical Analysis 1: Comparison: 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) vs Placebo; Logistic regression after multiple imputation. Analysis based on all available post-baseline body weight measurements (on-treatment (first intake of study drug until 28 days after last intake of study drug) and off-treatment), except those for participants who discontinued treatment early due to COVID-19. For these participants only on-treatment values were used; Test type: Other — Missing body weight measurements were multiply imputed using MMRM with treatment, gender, baseline body weight as factors. "Percentage change in body weight from baseline to Week 46" and "Body weight loss ≥ 5% at Week 46 (yes/no)" were derived per participant in each of the 1000 imputed datasets. Each dataset was analysed by a logistic regression. Multiple estimates from multiple imputation runs were summarised using Rubin's method; p = 0.0015, Regression, Logistic — P-value is considered nominal; Logistic regression with treatment group and gender as factors and baseline body weight as a continuous linear covariate; Odds Ratio (OR) = 3.28, 95% CI 2-sided [1.57 to 6.84] — Odds ratio is calculated as BI 456906 / Placebo
Statistical Analysis 2: Comparison: 2.4 mg BI 456906 - Planned Maintenance Treatment vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p < .0001, Regression, Logistic — P-value is considered nominal; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 8.83, 95% CI 2-sided [4.00 to 19.46] — Odds ratio is calculated as BI 456906 / Placebo
Statistical Analysis 3: Comparison: 3.6 mg BI 456906 - Planned Maintenance Treatment vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p < .0001, Regression, Logistic — P-value is considered nominal; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 7.48, 95% CI 2-sided [3.41 to 16.41] — Odds ratio is calculated as BI 456906 / Placebo
Statistical Analysis 4: Comparison: 4.8 mg BI 456906 - Planned Maintenance Treatment vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 2, analysis 1]; p < .0001, Regression, Logistic — P-value is considered nominal; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 10.77, 95% CI 2-sided [4.77 to 24.31] — Odds ratio is calculated as BI 456906 / Placebo

3. Secondary Outcome: Weight Loss of ≥ 10% of Baseline Weight at Week 46
Description: Weight loss of greater than or equal to 10 percent (≥10%) of baseline weight at Week 46 (yes/no), reported as percentage of participants who achieved a weight loss of ≥10% of baseline weight at Week 46. For analysis, all available post-baseline body weight measurements (on- and off-treatment) were used, except those for participants who discontinued treatment early due to COVID-19. For these participants only on-treatment values were used. Percentages were rounded to one decimal place.
Time Frame: At baseline and at Week 46.
Population: as for outcome 1
Measure: Number; unit: Percentage of participants
Arm/Group | 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) | 2.4 mg BI 456906 - Planned Maintenance Treatment | 3.6 mg BI 456906 - Planned Maintenance Treatment | 4.8 mg BI 456906 - Planned Maintenance Treatment | Placebo
Number analyzed (Participants) | 56 | 58 | 61 | 64 | 54
Percentage of participants | 33.9 | 65.5 | 65.6 | 68.8 | 11.1
Statistical Analysis 1: Comparison: 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other — Missing body weight measurements were multiply imputed using MMRM with treatment, gender, baseline body weight as factors. "Percentage change in body weight from baseline to Week 46" and "Body weight loss ≥ 10% at Week 46 (yes/no)" were derived per participant in each of the 1000 imputed datasets. Each dataset was analysed by a logistic regression. Multiple estimates from multiple imputation runs were summarised using Rubin's method; p = 0.0120, Regression, Logistic — P-value is considered nominal; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 3.22, 95% CI 2-sided [1.29 to 8.02] — Odds ratio is calculated as BI 456906 / Placebo
Statistical Analysis 2: Comparison: 2.4 mg BI 456906 - Planned Maintenance Treatment vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 3, analysis 1]; p < .0001, Regression, Logistic — P-value is considered nominal; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 10.62, 95% CI 2-sided [4.36 to 25.86] — Odds ratio is calculated as BI 456906 / Placebo
Statistical Analysis 3: Comparison: 3.6 mg BI 456906 - Planned Maintenance Treatment vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 3, analysis 1]; p < .0001, Regression, Logistic — P-value is considered nominal; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 9.78, 95% CI 2-sided [4.02 to 23.79] — Odds ratio is calculated as BI 456906 / Placebo
Statistical Analysis 4: Comparison: 4.8 mg BI 456906 - Planned Maintenance Treatment vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 3, analysis 1]; p < .0001, Regression, Logistic — P-value is considered nominal; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 14.50, 95% CI 2-sided [5.91 to 35.55] — Odds ratio is calculated as BI 456906 / Placebo

4. Secondary Outcome: Weight Loss of ≥ 15% of Baseline Weight at Week 46
Description: Weight loss of greater than or equal to 15 percent (≥15%) of baseline weight at Week 46 (yes/no), reported as percentage of participants who achieved a weight loss of ≥15% of baseline weight at Week 46. For analysis, all available post-baseline body weight measurements (on- and off-treatment) were used, except those for participants who discontinued treatment early due to COVID-19. For these participants only on-treatment values were used. Percentages were rounded to one decimal place.
Time Frame: At baseline and at Week 46.
Population: as for outcome 1
Measure: Number; unit: Percentage of particpants
Arm/Group | 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) | 2.4 mg BI 456906 - Planned Maintenance Treatment | 3.6 mg BI 456906 - Planned Maintenance Treatment | 4.8 mg BI 456906 - Planned Maintenance Treatment | Placebo
Number analyzed (Participants) | 56 | 58 | 61 | 64 | 54
Percentage of particpants | 12.5 | 37.9 | 45.9 | 54.7 | 5.6
Statistical Analysis 1: Comparison: 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other — Missing body weight measurements were multiply imputed using MMRM with treatment, gender, baseline body weight as factors. "Percentage change in body weight from baseline to Week 46" and "Body weight loss ≥ 15% at Week 46 (yes/no)" were derived per participant in each of the 1000 imputed datasets. Each dataset was analysed by a logistic regression. Multiple estimates from multiple imputation runs were summarised using Rubin's method; p = 0.2654, Regression, Logistic — P-value is considered nominal; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 2.13, 95% CI 2-sided [0.56 to 8.02] — Odds ratio is calculated as BI 456906 / Placebo
Statistical Analysis 2: Comparison: 2.4 mg BI 456906 - Planned Maintenance Treatment vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; p = 0.0002, Regression, Logistic — P-value is considered nominal; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 9.47, 95% CI 2-sided [2.89 to 30.95] — Odds ratio is calculated as BI 456906 / Placebo
Statistical Analysis 3: Comparison: 3.6 mg BI 456906 - Planned Maintenance Treatment vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; p < .0001, Regression, Logistic — P-value is considered nominal; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 11.79, 95% CI 2-sided [3.62 to 38.36] — Odds ratio is calculated as BI 456906 / Placebo
Statistical Analysis 4: Comparison: 4.8 mg BI 456906 - Planned Maintenance Treatment vs Placebo; [analysis description as in outcome 2, analysis 1]; Test type: Other — [test comment as in outcome 4, analysis 1]; p < .0001, Regression, Logistic — P-value is considered nominal; [statistical method as in outcome 2, analysis 1]; Odds Ratio (OR) = 21.02, 95% CI 2-sided [6.47 to 68.28] — Odds ratio is calculated as BI 456906 / Placebo

5. Secondary Outcome: Absolute Change in Body Weight From Baseline to Week 46
Description: Absolute change in body weight from baseline to Week 46 was modeled using a mixed model for repeated measures (MMRM) with fixed effects for baseline body weight as a continuous linear covariate, and treatment, gender, visit, treatment by visit interaction and baseline by visit interaction as factors, using visit (Week 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 28, 32, 36, 40, and 46) as repeated measures and an unstructured covariance matrix to model within subject measurements, adjusted mean (standard error) at Week 46 is reported. MMRM analysis was performed on the FAS, using planned maintenance treatment (dose assigned at randomisation) and including only on-treatment data, regardless of whether early treatment discontinuation was COVID-19 related.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 28, 32, 36, 40, and 46.
Population: Full analysis set (FAS, all randomised participants who received at least one dose of study treatment and who have analysable data for at least one efficacy endpoint), using planned maintenance treatment. Number of participants analysed = Participants with available data for the outcome measure.
Measure: Least Squares Mean (Standard Error); unit: Kilogram (kg)
Arm/Group | 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) | 2.4 mg BI 456906 - Planned Maintenance Treatment | 3.6 mg BI 456906 - Planned Maintenance Treatment | 4.8 mg BI 456906 - Planned Maintenance Treatment | Placebo
Number analyzed (Participants) | 75 | 78 | 76 | 76 | 76
Kilogram (kg) | -7.21 (1.06) | -14.75 (1.03) | -15.64 (1.04) | -18.47 (1.04) | -2.68 (1.04)
Statistical Analysis 1: Comparison: 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) vs Placebo; No formal hypotheses were tested; Test type: Other — [test comment as in outcome 1, analysis 6]; p = 0.0025, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger approximation was used to estimate the denominator degrees of freedom; Difference of adjusted means = -4.53, 95% CI 2-sided [-7.44 to -1.61], Standard Error of Mean 1.48 — Difference was calculated as BI 456906 - placebo
Statistical Analysis 2: Comparison: 2.4 mg BI 456906 - Planned Maintenance Treatment vs Placebo; No formal hypotheses were tested; Test type: Other — [test comment as in outcome 1, analysis 6]; p < .0001, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger approximation was used to estimate the denominator degrees of freedom; Difference of adjusted means = -12.07, 95% CI 2-sided [-14.94 to -9.19], Standard Error of Mean 1.46 — Difference was calculated as BI 456906 - placebo
Statistical Analysis 3: Comparison: 3.6 mg BI 456906 - Planned Maintenance Treatment vs Placebo; No formal hypotheses were tested; Test type: Other — [test comment as in outcome 1, analysis 6]; p < .0001, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger approximation was used to estimate the denominator degrees of freedom; Difference of adjusted means = -12.96, 95% CI 2-sided [-15.85 to -10.07], Standard Error of Mean 1.47 — Difference was calculated as BI 456906 - placebo at week 46
Statistical Analysis 4: Comparison: 4.8 mg BI 456906 - Planned Maintenance Treatment vs Placebo; No formal hypotheses were tested; Test type: Other — [test comment as in outcome 1, analysis 6]; p < .0001, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger approximation was used to estimate the denominator degrees of freedom; Difference of adjusted means = -15.78, 95% CI 2-sided [-18.67 to -12.90], Standard Error of Mean 1.47 — Difference was calculated as BI 456906 - placebo at week 46

6. Secondary Outcome: Absolute Change in Waist Circumference From Baseline to Week 46
Description: Absolute change in waist circumference from baseline to Week 46 was modeled using a mixed model for repeated measures (MMRM) with fixed effects for baseline waist circumference as a continuous linear covariate, and treatment, gender, visit, treatment by visit interaction and baseline by visit interaction as factors, using visit (Week 6, 12, 18, 24, 32, 40, and 46) as repeated measures and an unstructured covariance matrix to model within subject measurements, adjusted mean (standard error) at Week 46 is reported. MMRM analysis was performed on the FAS, using planned maintenance treatment (dose assigned at randomisation) and including only on-treatment data, regardless of whether early treatment discontinuation was COVID-19 related.
Time Frame: Baseline, Week 6, 12, 18, 24, 32, 40, and 46.
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Centimeter (cm)
Arm/Group | 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) | 2.4 mg BI 456906 - Planned Maintenance Treatment | 3.6 mg BI 456906 - Planned Maintenance Treatment | 4.8 mg BI 456906 - Planned Maintenance Treatment | Placebo
Number analyzed (Participants) | 71 | 71 | 74 | 75 | 72
Centimeter (cm) | -8.32 (1.22) | -14.99 (1.21) | -14.96 (1.19) | -16.01 (1.19) | -3.96 (1.20)
Statistical Analysis 1: Comparison: 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) vs Placebo; No formal hypotheses were tested; Test type: Other — MMRM with fixed effects for baseline waist circumference as a continuous linear covariate, and treatment, gender, visit, treatment by visit interaction and baseline by visit interaction as factors, using visit as repeated measures and an unstructured covariance matrix to model within subject measurements; p = 0.0116, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger approximation was used to estimate the denominator degrees of freedom; Difference of adjusted means = -4.36, 95% CI 2-sided [-7.74 to -0.98], Standard Error of Mean 1.71 — Difference was calculated as BI 456906 - placebo
Statistical Analysis 2: Comparison: 2.4 mg BI 456906 - Planned Maintenance Treatment vs Placebo; No formal hypotheses were tested; Test type: Other — [test comment as in outcome 6, analysis 1]; p < .0001, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger approximation was used to estimate the denominator degrees of freedom; Difference of adjusted means = -11.03, 95% CI 2-sided [-14.39 to -7.66], Standard Error of Mean 1.71 — Difference was calculated as BI 456906 - placebo
Statistical Analysis 3: Comparison: 3.6 mg BI 456906 - Planned Maintenance Treatment vs Placebo; No formal hypotheses were tested; Test type: Other — [test comment as in outcome 6, analysis 1]; p < .0001, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger approximation was used to estimate the denominator degrees of freedom; Difference of adjusted means = -11.00, 95% CI 2-sided [-14.33 to -7.67], Standard Error of Mean 1.69 — Difference was calculated as BI 456906 - placebo
Statistical Analysis 4: Comparison: 4.8 mg BI 456906 - Planned Maintenance Treatment vs Placebo; No formal hypotheses were tested; Test type: Other — [test comment as in outcome 6, analysis 1]; p < .0001, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger approximation was used to estimate the denominator degrees of freedom; Difference of adjusted means = -12.05, 95% CI 2-sided [-15.39 to -8.71], Standard Error of Mean 1.69 — Difference was calculated as BI 456906 - placebo

7. Secondary Outcome: Absolute Change in Systolic Blood Pressure From Baseline to Week 46
Description: Absolute change in systolic blood pressure from baseline to Week 46 was modeled using a mixed model for repeated measures (MMRM) with fixed effects for baseline systolic blood pressure as a continuous linear covariate, and treatment, gender, visit, treatment by visit interaction and baseline by visit interaction as factors, using visit Week 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 28, 32, 36, 40, and 46) as repeated measures and an unstructured covariance matrix to model within subject measurements, adjusted mean (standard error) at Week 46 is reported. MMRM analysis was performed on the FAS, using planned maintenance treatment (dose assigned at randomisation) and including only on-treatment data, regardless of whether early treatment discontinuation was COVID-19 related.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 28, 32, 36, 40, and 46.
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Millimeter of mercury (mmHg)
Arm/Group | 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) | 2.4 mg BI 456906 - Planned Maintenance Treatment | 3.6 mg BI 456906 - Planned Maintenance Treatment | 4.8 mg BI 456906 - Planned Maintenance Treatment | Placebo
Number analyzed (Participants) | 75 | 78 | 76 | 76 | 76
Millimeter of mercury (mmHg) | -6.19 (1.47) | -8.08 (1.48) | -8.66 (1.44) | -8.62 (1.46) | -2.46 (1.46)
Statistical Analysis 1: Comparison: 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) vs Placebo; No formal hypotheses were tested; Test type: Other — MMRM with fixed effects for baseline systolic blood pressure as a continuous linear covariate, and treatment, gender, visit, treatment by visit interaction and baseline by visit interaction as factors, using visit as repeated measures and an unstructured covariance matrix to model within subject measurements; p = 0.0733, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger approximation was used to estimate the denominator degrees of freedom; Difference of adjusted means = -3.73, 95% CI 2-sided [-7.82 to 0.35], Standard Error of Mean 2.08 — Difference was calculated as BI 456906 - placebo
Statistical Analysis 2: Comparison: 2.4 mg BI 456906 - Planned Maintenance Treatment vs Placebo; No formal hypotheses were tested; Test type: Other — [test comment as in outcome 7, analysis 1]; p < .0072, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger approximation was used to estimate the denominator degrees of freedom; Difference of adjusted means = -5.62, 95% CI 2-sided [-9.71 to 1.53], Standard Error of Mean 2.08 — Difference was calculated as BI 456906 - placebo
Statistical Analysis 3: Comparison: 3.6 mg BI 456906 - Planned Maintenance Treatment vs Placebo; No formal hypotheses were tested; Test type: Other — [test comment as in outcome 7, analysis 1]; p = 0.0027, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger approximation was used to estimate the denominator degrees of freedom; Difference of adjusted means = -6.20, 95% CI 2-sided [-10.23 to -2.17], Standard Error of Mean 2.05 — Difference was calculated as BI 456906 - placebo
Statistical Analysis 4: Comparison: 4.8 mg BI 456906 - Planned Maintenance Treatment vs Placebo; No formal hypotheses were tested; Test type: Other — [test comment as in outcome 7, analysis 1]; p = 0.0033, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger approximation was used to estimate the denominator degrees of freedom; Difference of adjusted means = -6.16, 95% CI 2-sided [-10.25 to -2.06], Standard Error of Mean 2.08 — Difference was calculated as BI 456906 - placebo

8. Secondary Outcome: Absolute Change in Diastolic Blood Pressure From Baseline to Week 46
Description: Absolute change in diastolic blood pressure from baseline to Week 46 was modeled using a mixed model for repeated measures (MMRM) with fixed effects for baseline diastolic blood pressure as a continuous linear covariate, and treatment, gender, visit, treatment by visit interaction and baseline by visit interaction as factors, using visit Week 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 28, 32, 36, 40, and 46) as repeated measures and an unstructured covariance matrix to model within subject measurements, adjusted mean (standard error) at Week 46 is reported. MMRM analysis was performed on the FAS, using planned maintenance treatment (dose assigned at randomisation) and including only on-treatment data, regardless of whether early treatment discontinuation was COVID-19 related.
Time Frame: Baseline, Week 2, 4, 6, 8, 10, 12, 14, 16, 18, 20, 24, 28, 32, 36, 40, and 46.
Population: as for outcome 5
Measure: Least Squares Mean (Standard Error); unit: Millimeter of mercury (mmHg)
Arm/Group | 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) | 2.4 mg BI 456906 - Planned Maintenance Treatment | 3.6 mg BI 456906 - Planned Maintenance Treatment | 4.8 mg BI 456906 - Planned Maintenance Treatment | Placebo
Number analyzed (Participants) | 75 | 78 | 76 | 76 | 76
Millimeter of mercury (mmHg) | -3.31 (0.90) | -4.36 (0.90) | -4.31 (0.87) | -4.80 (0.89) | -1.87 (0.89)
Statistical Analysis 1: Comparison: 0.6 mg BI 456906 - Planned Maintenance Treatment (Maintenance Dose Assigned at Randomisation) vs Placebo; No formal hypotheses were tested; Test type: Other — MMRM with fixed effects for baseline diastolic blood pressure as a continuous linear covariate, and treatment, gender, visit, treatment by visit interaction and baseline by visit interaction as factors, using visit as repeated measures and an unstructured covariance matrix to model within subject measurements; p = 0.2569, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger approximation was used to estimate the denominator degrees of freedom; Difference of adjusted means = -1.44, 95% CI 2-sided [-3.92 to 1.05], Standard Error of Mean 1.26 — Difference was calculated as BI 456906 - placebo
Statistical Analysis 2: Comparison: 2.4 mg BI 456906 - Planned Maintenance Treatment vs Placebo; No formal hypotheses were tested; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.0495, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger approximation was used to estimate the denominator degrees of freedom; Difference of adjusted means = -2.49, 95% CI 2-sided [-4.97 to -0.00], Standard Error of Mean 1.26 — Difference was calculated as BI 456906 - placebo
Statistical Analysis 3: Comparison: 3.6 mg BI 456906 - Planned Maintenance Treatment vs Placebo; No formal hypotheses were tested; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.0506, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger approximation was used to estimate the denominator degrees of freedom; Difference of adjusted means = -2.44, 95% CI 2-sided [-4.90 to 0.01], Standard Error of Mean 1.24 — Difference was calculated as BI 456906 -placebo
Statistical Analysis 4: Comparison: 4.8 mg BI 456906 - Planned Maintenance Treatment vs Placebo; No formal hypotheses were tested; Test type: Other — [test comment as in outcome 8, analysis 1]; p = 0.0202, Mixed Models Analysis — P-value is considered nominal; Kenward-Roger approximation was used to estimate the denominator degrees of freedom; Difference of adjusted means = -2.93, 95% CI 2-sided [-5.40 to -0.46], Standard Error of Mean 1.25 — Difference was calculated as BI 456906 - placebo

ADVERSE EVENTS:
Time Frame: From first drug administration until last drug administration, plus 28 days residual effect period (REP), up to 360 days.
Description: Safety analysis was performed on the treated set (TS) according to actual maintenance treatment (defined as the actual dose participants received during the dose maintenance phase, or as the next planned maintenance dose up from the last dose taken prior to treatment discontinuation).
  Treated Set (TS): All randomised participants who received at least one dose of study treatment.
Groups:
- 0.6 mg BI 456906 - Actual Maintenance Treatment: Participants with obesity or overweight were administered a solution for injection of BI 456906, by a weekly subcutaneous injection of two syringes (0.5 mL filling volume per syringe) on the same injection day, of 0.3 mg on Week 1 and 2, and 0.6 mg on Week 3 to Week 20 (dose escalation phase, with fixed dose escalation from Week 1 to Week 10 and flexible dose escalation from Week 11 to Week 20).
  From Week 21 to Week 46 (maintenance dosing phase) participants stayed on the dose of 0.6 mg BI 456906.
  Participant not tolerating the assigned dose escalation schedule due to gastrointestinal adverse events had the option of dose adjustment during the flexible part of the dose escalation phase (Week 11 - 20) which could lead to a maintenance dose lower than the dose the participant was randomised to.
- 2.4 mg BI 456906 - Actual Maintenance Treatment: Participants with obesity or overweight were administered a solution for injection of BI 456906, by a weekly subcutaneous injection of two syringes (0.5 mL filling volume per syringe) on the same injection day, of 0.3 mg on Week 1 and Week 2, 0.6 mg on Week 3 and Week 4, 0.9 mg on Week 5 and Week 6, 1.2 mg on Week 7 to Week 10, 1.8 mg on Week 11 to Week 14 and 2.4 mg on Week 15 to Week 20 (dose escalation phase, with fixed dose escalation from Week 1 to Week 10 and flexible dose escalation from Week 11 to Week 20). From Week 21 to Week 46 (maintenance dosing phase) participants stayed on the dose of 2.4 mg BI 456906.
  Participant not tolerating the assigned dose escalation schedule due to gastrointestinal adverse events had the option of dose adjustment during the flexible part of the dose escalation phase (Week 11 - 20) which could lead to a maintenance dose lower than the dose the participant was randomised to.
- 3.6 mg BI 456906 - Actual Maintenance Treatment: Participants with obesity or overweight were administered a solution for injection of BI 456906, by a weekly subcutaneous injection of two syringes (0.5 mL filling volume per syringe) on the same injection day, of 0.3 mg on Week 1 and Week 2, 0.6 mg on Week 3 and Week 4, 0.9 mg on Week 5 and Week 6, 1.2 mg on Week 7 to Week 10, 1.8 mg on Week 11 and Week 12, 2.4 mg on Week 13 and Week 14, 3.0 mg on Week 15 and Week 16, and 3.6 mg on Week 17 to Week 20 (dose escalation phase, with fixed dose escalation from Week 1 to Week 10 and flexible dose escalation from Week 11 to Week 20). From Week 21 to Week 46 (maintenance dosing phase) participants stayed on the dose of 3.6 mg BI 456906.
  Participant not tolerating the assigned dose escalation schedule due to gastrointestinal adverse events had the option of dose adjustment during the flexible part of the dose escalation phase (Week 11 - 20) which could lead to a maintenance dose lower than the dose the participant was randomised to.
- 4.8 mg BI 456906 - Actual Maintenance Treatment: Participants with obesity or overweight were administered a solution for injection of BI 456906, by a weekly subcutaneous injection of two syringes (0.5 mL filling volume per syringe) on the same injection day, of 0.3 mg on Week 1 and Week 2, 0.6 mg on Week 3 and Week 4, 0.9 mg on Week 5 and Week 6, 1.2 mg on Week 7 and Week 8, 1.8 mg on Week 9 and Week 10, 2.4 mg on Week 11 and Week 12, 3.3 mg on Week 13 and Week 14, 4.2 mg on Week 15 and Week 16, and 4.8 mg on Week 17 to Week 20 (dose escalation phase, with fixed dose escalation from Week 1 to Week 10 and flexible dose escalation from Week 11 to Week 20). From Week 21 to Week 46 (maintenance dosing phase) participants stayed on the dose of 4.8 mg BI 456906.
  Participant not tolerating the assigned dose escalation schedule due to gastrointestinal adverse events had the option of dose adjustment during the flexible part of the dose escalation phase (Week 11 - 20) which could lead to a maintenance dose lower than the dose the participant was randomised to.
Arm/Group | 0.6 mg BI 456906 - Actual Maintenance Treatment | 2.4 mg BI 456906 - Actual Maintenance Treatment | 3.6 mg BI 456906 - Actual Maintenance Treatment | 4.8 mg BI 456906 - Actual Maintenance Treatment | Placebo
All-Cause Mortality (participants affected / at risk) | 0/92 | 0/92 | 0/71 | 0/54 | 0/77
Serious Adverse Events (participants affected / at risk) | 2/92 | 3/92 | 4/71 | 4/54 | 5/77
Other Adverse Events (participants affected / at risk) | 70/92 | 79/92 | 64/71 | 46/54 | 48/77
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | 0.6 mg BI 456906 - Actual Maintenance Treatment (N=92) | 2.4 mg BI 456906 - Actual Maintenance Treatment (N=92) | 3.6 mg BI 456906 - Actual Maintenance Treatment (N=71) | 4.8 mg BI 456906 - Actual Maintenance Treatment (N=54) | Placebo (N=77)
Deafness (Ear and labyrinth disorders) | 0 | 1 | 0 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 0 | 0 | 1 | 0
COVID-19 pneumonia (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Tonsillitis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Tooth abscess (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Incisional hernia (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Bowen's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0 | 0
Glioblastoma multiforme (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1 | 0
Intraductal proliferative breast lesion (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0 | 0
Renal failure (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Endometrial hyperplasia (Reproductive system and breast disorders) | 0 | 0 | 0 | 0 | 1
Uterine prolapse (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Pulmonary congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Angioedema (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 0.6 mg BI 456906 - Actual Maintenance Treatment (N=92) | 2.4 mg BI 456906 - Actual Maintenance Treatment (N=92) | 3.6 mg BI 456906 - Actual Maintenance Treatment (N=71) | 4.8 mg BI 456906 - Actual Maintenance Treatment (N=54) | Placebo (N=77)
Abdominal distension (Gastrointestinal disorders) | 4 | 4 | 7 | 3 | 3
Abdominal pain (Gastrointestinal disorders) | 4 | 10 | 5 | 3 | 1
Abdominal pain upper (Gastrointestinal disorders) | 3 | 5 | 8 | 2 | 1
Constipation (Gastrointestinal disorders) | 11 | 19 | 22 | 13 | 4
Diarrhoea (Gastrointestinal disorders) | 22 | 21 | 17 | 9 | 8
Dyspepsia (Gastrointestinal disorders) | 7 | 9 | 8 | 7 | 3
Eructation (Gastrointestinal disorders) | 4 | 6 | 5 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 7 | 10 | 5 | 3
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 3 | 1
Nausea (Gastrointestinal disorders) | 36 | 60 | 45 | 32 | 15
Vomiting (Gastrointestinal disorders) | 13 | 28 | 28 | 13 | 4
Fatigue (General disorders) | 6 | 5 | 13 | 5 | 6
Injection site bruising (General disorders) | 3 | 3 | 2 | 3 | 4
COVID-19 (Infections and infestations) | 18 | 11 | 17 | 7 | 17
Nasopharyngitis (Infections and infestations) | 8 | 5 | 6 | 3 | 7
Upper respiratory tract infection (Infections and infestations) | 2 | 1 | 5 | 4 | 3
Urinary tract infection (Infections and infestations) | 4 | 2 | 6 | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 11 | 10 | 16 | 3 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 10 | 3 | 8 | 2 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 7 | 2 | 4 | 2 | 3
Dizziness (Nervous system disorders) | 1 | 8 | 10 | 4 | 2
Headache (Nervous system disorders) | 8 | 7 | 10 | 5 | 6
Insomnia (Psychiatric disorders) | 3 | 5 | 1 | 1 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 4 | 0 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.

DOCUMENTS (2):
  • Study Protocol (2022-04-29): https://cdn.clinicaltrials.gov/large-docs/77/NCT04667377/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-08): https://cdn.clinicaltrials.gov/large-docs/77/NCT04667377/SAP_001.pdf